CLINICAL TRIAL: NCT01342835
Title: Postoperative Analgesia in Children After Propofol Anesthesia
Acronym: propan
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinical Centre of Kosova (Other)
Responsible Party: Antigona Hasani, UCCK
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCCK-55; RAA12 (Registry Identifier: RAA12)
Record Dates: First submitted 2011-04-20; First posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2010-09

CONDITIONS: Postoperative Pain
Keywords: propofol; sevoflurane; postoperative pain; children
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug: propofol (Active Comparator): Drug:Propofol and sevoflurane The induction dose of propofol is 3-5 mg/kg-1 (mean induction dose: 4 mg/kg-1) follow by propofol infusion (12 mg/kg/h-1 for the first 10 min of general anesthesia, 9 mg/kg/h-1 for another 10 min, and 6 mg/kg/h-1 thereafter; mean maintenance dose: 9 mg/kg/h-1) and a 50:50 mixture of N2O and O2.
  Interventions: Drug: Propofol
- Sevoflurane group:sevoflurane (Active Comparator): Drug:Sevoflurane and Propofol Mask induction is perform with sevoflurane (4-6%) follow by 1.5-2% sevoflurane in a 50:50 mixture of N2O and O2.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The induction dose of propofol is 3-5 mg/kg-1 (mean induction dose: 4 mg/kg-1) follow by propofol infusion (12 mg/kg/h-1 for the first 10 min of general anesthesia, 9 mg/kg/h-1 for another 10 min, and 6 mg/kg/h-1 thereafter; mean maintenance dose: 9 mg/kg/h-1) and a 50:50 mixture of N2O and O2.
  Other Names: Diprivan; Sevorane

SUMMARY:
The investigators hypothesize that patients anesthetized with sevoflurane have more pain, postoperatively, than those anesthetized with propofol.

DETAILED DESCRIPTION:
In a randomize, prospective, double-blind study, the subjects are 100 premedicated children, aged 3 to 6 years, who undergo one type of surgical procedure, hernia repair surgery. Anesthesia is maintains with propofol anesthesia (group P, n=50) or with sevoflurane anesthesia (group S, n=50). and fentanyl administered during surgery. Faces Pain Scale (FPS) is use to assess pain severity.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 3- 6 years old
* Patient is scheduled for hernia repair surgery at University Clinical center of Kosovo Patients is ASA I/II Patient meets criteria to receive either propofol or sevoflurane anesthesia Patient's parent/guardian provides written consent

Exclusion Criteria:

* allergy to any of the drugs
* preoperative anxiety
* postoperative agitation
* ASA physical status >II

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 120 minutes
  The Faces Pain Scale (FPS) (from five face drawings: 0 = no pain, 5 = extreme pain) is used to assess pain severity

SECONDARY OUTCOMES:
recovery time | 120 minutes
  Recovery time, defined as the time until eye opening on command or the time of first response to command after anesthesia
adverse effects | 0-120 minutes
  Adverse effects during the surgery and after recovery: hypotension, bradicardia, intense coughing, hypersalivation and laryngospasm, nausea, and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Antigona Hasani, MD,MSC, Principal Investigator — University Clinical Centre of Kosova
Locations (1):
- University Clinical Center of Kosovo, Pristina, Kosovo, Serbia